CLINICAL TRIAL: NCT01273129
Title: Surgery as a Treatment for Medically Intractable Epilepsy
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110051; 11-N-0051
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09-05

CONDITIONS: Epilepsy; Epilepsy, Temporal Lobe; Partial Epilepsy
Keywords: Neurosurgery; Childhood Epilepsy; Epilepsy; Frontal Lobe Epilepsy; Temporal Lobe Epilepsy; Natural History
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Epilepsies, Partial; Epilepsy, Frontal Lobe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients 8 years and older whose seizures are uncontrollable with medication may participate in this study as well as patients with tumor related epilepsy in whom invasive monitoring is indicated.

SUMMARY:
Background:

- Drug resistant epilepsy is the term used to describe epilepsy that cannot be controlled by medication. Many people whose seizures do not respond to medication will respond to surgical treatment, relieving seizures completely or almost completely in one-half to two-thirds of patients who qualify for surgery. The tests and surgery performed as part of this treatment are not experimental, but researchers are interested in using the data collected as part of routine standard epilepsy care to better understand epilepsy and its treatment.

Objectives:

- To use surgery as a treatment for drug resistant epilepsy in children and adults.

Eligibility:

- Children and adults at least 8 years of age who have simple or complex partial seizures (seizures that come from one area of the brain) that have not responded to medication, and who are willing to have brain surgery to treat their medically intractable epilepsy.

Design:

* Participants will be screened with a medical history, physical examination, and neurological examination. Imaging studies, including magnetic resonance imaging and computer-assisted tomography (CT), may also be conducted as part of the screening. Participants who do not need surgery or whose epilepsy cannot be treated surgically will follow up with a primary care physician or neurologist and will not need to return to the National Institutes of Health for this study.
* Prior to the surgery, participants will have the following procedures to provide information on the correct surgical approach.
* Video electroencephalography monitoring to measure brain activity during normal activities within a 24-hour period. Three to four 15-minute breaks are allowed within this period.
* Electrodes placed directly in the brain or on the surface of the brain to measure brain activities and determine the part of the brain that is responsible for the seizures (seizure focus).
* Participants will have a surgical procedure at the site of their seizure focus. Brain lesions, abnormal blood vessels, tumors, infections, or other areas of brain abnormality will be either removed or treated in a way that will stop or help prevent the spread of seizures without affecting irreplaceable brain functions, such as the ability to speak, understand, move, feel, or see.
* Participants will return for outpatient visits and brain imaging studies 2 months, 1 year, and 2 years after surgery.

DETAILED DESCRIPTION:
Objective

This protocol is being performed to collect prospective data on patients who receive standard of care treatment for drug resistant epilepsy and to follow the natural history of patients receiving epilepsy surgery, to investigate neurophysiological correlates of human cognitive function, to provide invasive monitoring for patients with tumor related epilepsy. Any treatment under this protocol will be based on the current standard of care for epilepsy surgery.

Study Population

Patients 8 years and older whose seizures are uncontrollable with medication may participate in this study as well as patients with tumor related epilepsy in whom invasive monitoring is indicated.

Study Design

Patients will be screened by study neurologists to confirm their diagnosis of drug resistant epilepsy. Patients that do not have a confirmed diagnosis of drug resistant epilepsy will be offered further evaluation in protocol 18-N-0066, Investigating Epilepsy: Screening, Evaluation and Treatment. Patients confirmed to have drug resistant epilepsy will be offered standard invasive and non-invasive diagnostic and surgical procedures. Diagnostic invasive monitoring with intracranial electrodes for further localization of their seizure focus may be required. The ultimate goal is to surgically remove or modify the epileptic focus. Standard procedures to be performed are 1) anterior temporal lobectomy or 2) amygdalohippocampectomy for temporal lobe epilepsy, 3) focal cortical resection for epilepsy that arises outside the temporal lobe, 4) removal of brain lesions causing epilepsy, 5) multiple subpial transection, and 6) placement of neurostimulator devices. These procedures are all FDA approved standard of care for treatment of drug resistant epilepsy.

In patients in whom invasive monitoring is medically necessary, neurophysiologic activity during cognitive tasks will be captured from intracranial surface and depth electrodes. Analysis will focus on the role of neuronal firing and aggregate neural activity 1) during cognitive function, 2) in other states such as wakefulness and sleep, and 3) during periods of time surrounding seizure activity.

Drug Resistant Epilepsy

Patients with drug resistant epilepsy will be followed for three months after the surgical procedure and will receive standard neurological examinations and MRI evaluation of the brain. Participants in this protocol will be evaluated for potential eligibility for other NINDS clinical trials.

Tumor Related epilepsy

Patients with tumor related epilepsy will be enrolled in this protocol because of clinical indications arising from participation in a separate protocol, 16-N-0041 Tumor Related Epilepsy. Patients will complete participation after the three-month post-op visit.

Outcome Measures

By providing standard care treatment for patients with drug resistant epilepsy, this protocol allows for descriptive and/or correlational studies based on the data collected through clinical care of these patients including neurophysiological correlates of cognitive function and studies of tissue sample acquired during surgery. Outcomes for patients with tumor related epilepsy will be assessed under a separate protocol, 16-N-0041, Tumor Related Epilepsy.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, candidates must:

1. Be 8 years of age or older with drug resistant epilepsy or tumor related epilepsy.

EXCLUSION CRITERIA:

Candidates will be excluded if they:

1. Are unable or unwilling to give informed consent, or have a parent able to provide informed consent if a minor, to the research procedures.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 8 years and older whose seizures are uncontrollable with medication may participate in this study as well as patients with tumor related epilepsy in whom invasive monitoring is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-03-21 (Actual)

PRIMARY OUTCOMES:
Descriptive and/or correlational studies | 1 year
  By providing standard care treatment for patients with drug resistant epilepsy, this protocol allows for descriptive and/or correlational studies based on the data collected through clinical care of these patients including neurophysiological correlates of cognitive function and studies of tissue sample acquired during surgery. Outcomes for patients with tumor related epilepsy will be assessed under a separate protocol, 16-N-0041, Tumor Related Epilepsy.

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. we will share all IPD that results in a publication on a public repository, as required by most journals. the data will be de-identified and anonymized.

REFERENCES:
- [Derived] Chittajallu R, Auville K, Mahadevan V, Lai M, Hunt S, Calvigioni D, Pelkey KA, Zaghloul KA, McBain CJ. Activity-dependent tuning of intrinsic excitability in mouse and human neurogliaform cells. Elife. 2020 Jun 4;9:e57571. doi: 10.7554/eLife.57571. PMID 32496194
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-N-0051.html